CLINICAL TRIAL: NCT03059511
Title: Pharmacokinetics of Nalbuphine After Intravenous and Intranasal Administration in Infants: A Single Center, Open-label, Prospective Study
Brief Title: Pharmacokinetics of Nalbuphine After Intravenous and Intranasal Administration in Infants
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: We conclude that the doses we administered were safe, but too low. We plan to continue the study with higher doses (0.1 mg/kg iv and 0.2 mg/kg intranasal).
Sponsor: University Children's Hospital, Zurich (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PK_Nalbuphin_iv_intranasal
Record Dates: First submitted 2017-02-06; First posted 2017-02-23 (Actual); Last update posted 2021-12-14 (Actual); Status verified 2021-12

CONDITIONS: Pharmacokinetic
MeSH Terms: interventions — Nalbuphine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- intravenous (Active Comparator): single iv application of nalbuphine 0.05mg/kg
  Interventions: Drug: Nalbuphine
- intranasal (Active Comparator): single intranasal application of nalbuphine 0.1mg/kg in infants.
  Interventions: Drug: Nalbuphine

INTERVENTIONS:
Drug: Nalbuphine — Opioid Pain Medicine

SUMMARY:
To assess pharmacokinetics parameters for nalbuphine after intravenous and intranasal administration in infants. Also effect on pain score: Neonatal Infant Pain Score (NIPS) and safety will be evaluated with summary of Adverse Events.

Inclusion criteria are: Infants 29 days-3 months, minimum Body weight 3.0 kg, Indications: septical work up.

Exclusion criteria are: Infants who were born prematurely (before 37 weeks gestation), known kidney or liver disease, known chronic illness.

ELIGIBILITY:
Inclusion Criteria:

* Infants 29 days-3 months
* Minimum Body weight 3.0 kg
* Indications: septical work up
* Parent has been informed about the study and has signed Informed Consent Form

Exclusion Criteria:

* Infants who were born prematurely (before 37 weeks gestation)
* Known kidney or liver disease
* Known chronic illness
* Documented previous adverse reaction to nalbuphine
* Treatment with a depressant drug within 5 days prior to study
* Epistaxis, nose trauma (only for the intranasal application)
* Barriere of language

Ages: 29 Days to 3 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 51 (Actual)
Dates: Start 2017-03-03 (Actual); Primary Completion 2018-01-10 (Actual); Study Completion 2018-01-10 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics (Area under the plasma concentration-time) | One Visit = approximately 6 hours
  Area under the plasma concentration-time from the first to the last sample
Pharmacokinetics (Maximum Plasma concentration) | One Visit = approximately 6 hours
  Maximum Plasma concentration
Pharmacokinetics (Time to reach Maximum Plasma concentration) | One Visit = approximately 6 hours
  Time to reach Maximum Plasma concentration
Pharmacokinetics (Half-life time) | One Visit = approximately 6 hours
  Half-life time
Pharmacokinetics (Bioavailability of Nalbuphine intranasal) | One Visit = approximately 6 hours
  Bioavailability of Nalbuphine intranasal

SECONDARY OUTCOMES:
Effect on pain (Neonatal Infant Pain Score) | One Visit = approximately 6 hours
  Effect on pain score: NIPS (Neonatal Infant Pain Score)
Adverse Events | One Visit = approximately 6 hours
  Safety will be evaluated with summary of Adverse Events

CONTACTS AND LOCATIONS:
Overall Officials: Eva Berger, Dr, Principal Investigator — Chlidrens Hospital Zurich
Locations (1):
- Childens Hospital Zurich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
if someone ask for IPD

REFERENCES:
- [Derived] Pfiffner M, Gotta V, Pfister M, Vonbach P, Berger-Olah E. Pharmacokinetics and tolerability of intranasal or intravenous administration of nalbuphine in infants. Arch Dis Child. 2023 Jan;108(1):56-61. doi: 10.1136/archdischild-2022-323807. Epub 2022 Sep 13. PMID 36100355